CLINICAL TRIAL: NCT02573454
Title: Prosocial Exercise: Does Exercising for Charity Result in Greater Well-Being and Physical Activity?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Mark Beauchamp, Dr. Mark Beauchamp, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H14-03018
Record Dates: First submitted 2015-10-07; First posted 2015-10-09 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prosocial Exercise (Experimental): Participants are provided with the intervention (App Assignment). In this arm, the participants are randomly assigned to the Prosocial Exercise group use a GPS exercise app named Charity Miles, in which users can earn donations for charities based on the miles they walk or run (approximately 25 cents for every mile).
  Interventions: Behavioral: App assignment
- Personal Exercise (Active Comparator): Participants are provided with the intervention (App Assignment). In this arm, the participants are randomly assigned to the Personal Exercise group use a traditional GPS exercise app named Nike + Running, in which users can track the mileage that they walk or run (i.e., there is no opportunity to earn donations for charity through exercise behaviour).
  Interventions: Behavioral: App assignment

INTERVENTIONS:
Behavioral: App assignment — Under-active undergraduates are assigned to use a GPS exercise app that is prosocial (i.e., allows the user to raise money for charities) or personal (does not allow the user to raise money for charities) in nature

SUMMARY:
The purpose of this study is to determine whether prosocial exercise (exercising for the benefit of others) results in greater well-being and physical activity when compared to personal exercise (exercising without attempting to benefit others). Participants will be randomly assigned to utilize one of two exercise apps for a two week period: Charity Miles, which allows users to donate money to charities based on exercise participation, or Nike+ Running, which is a standard GPS exercise app. Participants will be provided with questionnaires at pre- and post-test, at a 4 week-follow-up, and immediately before and after each use of the app.

DETAILED DESCRIPTION:
Physical inactivity is a prevalent problem, with few Canadians active enough to accrue the health-related benefits associated with exercise. In response to ineffective means of physical activity promotion efforts, recent work suggests focusing on well-being as an outcome of exercise to better promote such behaviour.

Well-being is often conceptualized from two separate fields of study: hedonia and eudaimonia. Hedonia is concerned with the experience of pleasure and the avoidance of pain and is often equated to happiness. Conversely, eudaimonia is associated with more existential concerns and is sometimes equated with 'personal meaning'.

While hedonic well-being has been reliably linked to increased physical activity behaviour, less is understood about the possible effects of eudaimonic well-being on exercise engagement. As such, research should work towards developing a greater understanding of the relationship between well-being and physical activity. In doing so, research may be able to ascertain whether the experience of both hedonic and eudaimonic well-being is effective in increasing exercise engagement.

One particular behaviour that has been reliably linked to well-being is prosocial behaviour, or behaviour undertaken voluntarily with the aim of aiding or benefitting others. In particular, a wide variety of research has established a link between well-being and prosocial behaviours including volunteering and prosocial spending. Furthermore, engaging in prosocial behaviour has been identified as an effective means of motivating individuals and increasing performance.

As prosocial behaviour has been linked to increased hedonic and eudaimonic well-being, and as prosocial motivation has been identified as a powerful means of behaviour change, prosocial exercise, or engaging in physical activity to benefit others, may produce increases in well-being and future physical activity behaviour. As prosocial exercise is a common and popular activity (e.g., engaging in charity runs such as Run for the Cure or Relay for Life), research should work to ascertain whether increased well-being is related to prosocial exercise, and whether this association results in increased exercise behaviour.

In order to test this, students will be recruited to take part in a two-week experiment, whereby half of the students will be randomly assigned to a prosocial exercise condition (and use the prosocial exercise app, 'Charity Miles'), and half will be randomly assigned to a personal exercise condition (and utilize a standard exercise app, Nike+ Running). Participants' eudaimonic and hedonic well-being and exercise behaviour will be assessed at baseline and two weeks following, as well as before and after each use of the exercise app. It is hypothesized that the participants in the prosocial exercise condition will report greater exercise engagement compared to participants in the standard condition, and that this relationship will be mediated by hedonic and eudaimonic well-being.

ELIGIBILITY:
Inclusion Criteria:

* able to read and write English,
* undergraduate student at UBC,
* owns a smart phone (i.e., android or iPhone), and
* participates in a maximum of three 30 minute sessions of moderate-vigorous activity per week.

Exclusion Criteria:

* individuals not cleared for physical activity engagement (i.e., those that do not pass the Physical Activity Readiness Questionnaire Plus (PAR-Q+) and do not obtain a doctor's approval).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Moderate-Vigorous Physical Activity assessed by the Godin's Leisure Time Exercise Questionnaire (GLTEQ) | Pre-test, 2-weeks post, 6-weeks post
  A modified version of the Godin's Leisure Time Exercise Questionnaire (GLTEQ; Godin & Shephard, 1985) is employed

CONTACTS AND LOCATIONS:
Overall Officials: Mark Beauchamp, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Colley RC, Garriguet D, Janssen I, Craig CL, Clarke J, Tremblay MS. Physical activity of Canadian adults: accelerometer results from the 2007 to 2009 Canadian Health Measures Survey. Health Rep. 2011 Mar;22(1):7-14. PMID 21510585
- [Background] Segar ML, Eccles JS, Richardson CR. Rebranding exercise: closing the gap between values and behavior. Int J Behav Nutr Phys Act. 2011 Aug 31;8:94. doi: 10.1186/1479-5868-8-94. PMID 21884579
- [Background] Segar ML, Richardson CR. Prescribing pleasure and meaning: cultivating walking motivation and maintenance. Am J Prev Med. 2014 Dec;47(6):838-41. doi: 10.1016/j.amepre.2014.07.001. Epub 2014 Aug 26. No abstract available. PMID 25172091
- [Background] Ryan RM, Deci EL. On happiness and human potentials: a review of research on hedonic and eudaimonic well-being. Annu Rev Psychol. 2001;52:141-66. doi: 10.1146/annurev.psych.52.1.141. PMID 11148302
- [Background] Rhodes RE, Fiala B, Conner M. A review and meta-analysis of affective judgments and physical activity in adult populations. Ann Behav Med. 2009 Dec;38(3):180-204. doi: 10.1007/s12160-009-9147-y. PMID 20082164
- [Background] Bierhoff, H. W. (2005). Prosocial behaviour. New York: Psychology Press.
- [Background] Thoits PA, Hewitt LN. Volunteer work and well-being. J Health Soc Behav. 2001 Jun;42(2):115-31. PMID 11467248
- [Background] Dunn EW, Aknin LB, Norton MI. Spending money on others promotes happiness. Science. 2008 Mar 21;319(5870):1687-8. doi: 10.1126/science.1150952. PMID 18356530
- [Background] Grant, A. M., Campbell, E. M., Chen, G., Cottone, K., Lapedis, D., & Lee, K. (2007). Impact and the art of motivation maintenance: The effects of contact with beneficiaries on persistence behavior. Organizational Behavior and Human Decision Processes, 103(1), 53-67.